CLINICAL TRIAL: NCT03707912
Title: Multicentre Double-blind Placebo-controlled Parallel Group Randomized Clinical Trial of Efficacy and Safety of Anaferon in the Treatment of Acute Respiratory Viral Infections
Brief Title: Clinical Trial of Efficacy and Safety of Anaferon in the Treatment of Acute Respiratory Viral Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-AN-005
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Acute Respiratory Viral Infections
MeSH Terms: interventions — anaferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaferon (Experimental): 1 tablet per administration. Day 1: 1 tablet every 30 minutes for the first 2 hours, followed by 3 more tablets taken at regular intervals through the rest of the day.
  Days 2-5: 1 tablet 3 times a day. The drug is taken out of the meal (in the interval between meals or 15-30 minutes before eating), keep the tablet in the mouth, without swallowing, until completely dissolved.
  Interventions: Drug: Anaferon
- Placebo (Placebo Comparator): Placebo using Anaferon regimen until the end of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anaferon — Oral administration.
  Arms: Anaferon
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
Purpose of the study:

• To obtain additional data on the efficacy and safety of Anaferon in the treatment of acute respiratory viral infections.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, parallel-group randomized trial.

The study will enroll patients of either gender aged 18-70 years old with clinical manifestations of ARVI within the first day after the onset of the disease. Signed information sheet for patient will be obtained from all participants prior to the screening procedures. Medical history, concomitant medication, thermometry, patient examination by a doctor, assessment of ARVI symptoms severity will be performed at screening visit.

The nasopharyngeal swabs will be performed for Real-time reverse transcription polymerase chain reaction (PCR) assay to confirm viral etiology of ARVI and to verify respiratory viruses prior to the therapy.

If a patient meets all inclusion criteria and does not have any exclusion criteria, at Visit 1 (Day 1) he/she will be randomized into one of two groups: the 1st group patients will take Anaferon according to the dosage regimen until the end of the study; the 2nd group patients will take Placebo according to Anaferon dosage regimen until the end of the study.

The patients will be provided with a patient diary (paper or electronic) where daily they will record axillary body temperature (using a Geratherm Classic thermometer) and each ARVI symptom severity twice a day (in the morning and in the evening). In addition, antipyretic administration (if applicable) as well as any possible worsening of the patient's condition (if applicable, for safety evaluation/AEs documentation) will also be recorded in a patient diary. An investigator will provide the instructions on filling out the diary and will help the patient to make first records of ARVI symptom severity and body temperature in the diary.

Patients are observed up for 7 days (screening, randomization - 1 day, study therapy - 5 days, follow-up period - 2 days). During treatment and follow-up period two visits are scheduled (at home or at the study site) on days 5 (Visit 2) and day 7 (Visit 3). At Visits 2 and 3, the investigator will carry out physical examination, record dynamics of ARVI symptoms and concomitant therapy and check patient diaries.

Treatment compliance will be evaluated at Visit 3. During the study, symptomatic therapy and therapy for underlying chronic conditions are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender aged 18-70 years.
2. Diagnosis of acute respiratory viral infection (ARVI) based on medical examination: axillary temperature ≥ 37,8 ° C at examination + non-specific/flu-like symptom score ≥4, nasal/throat/chest symptom score ≥2.
3. The first 24 hours after ARVI onset.
4. Seasonal rise in ARVI incidence.
5. Patients giving their consent to use reliable contraception during the study.
6. Signed patient information sheet (informed consent form).

Exclusion Criteria:

1. Suspected pneumonia, bacterial infection (including otitis media, sinuitis, urinary tract infection, meningitis, sepsis, etc.), requiring the administration of antibacterial drugs from the first day of the disease.
2. Suspected initial manifestations of diseases with symptoms similar to ARVI at onset (other infectious diseases, flu-like syndrome at the onset of systemic diseases of connective tissue, oncohaematological and other diseases).
3. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
4. Subjects requiring concurrent antiviral products forbidden by the study.
5. Medical history of primary and secondary immunodeficiency.
6. Oncologic conditions /suspected oncologic conditions.
7. Aggravation or decompensation of chronic diseases affecting a patient's ability to participate in the clinical trial.
8. Impaired glucose tolerance, diabetes mellitus.
9. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
10. Allergy/ hypersensitivity to any component of the study drug.
11. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial.
12. Consumption of narcotics, alcohol > 2 alcohol units per day, mental diseases.
13. Course administration of the drug products specified in the section "Prohibited Concomitant Therapy" within two weeks prior to inclusion in the study.
14. Patients who will not fulfill the requirements during the study or follow the order of administration of the studied drug products, from the Investigator's point of view.
15. Participation in other clinical trials for 3 months prior to enrollment in this study.
16. Patients who are related to any of the on-site research personnel directly involved in the study or are an immediate relative of the investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
17. Patients who work for OOO "NPF "Materia Medica Holding" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Russia (19):
  - Regional State Budgetary Healthcare Institution "City Hospital No. 5, Barnaul", Barnaul
  - Non-governmental health care institution "Road Clinical Hospital at Chelyabinsk station JSC" Russian Railways ", Chelyabinsk
  - Kazan State Medical University, Kazan'
  - Krasnogorsk city hospital №1, Krasnogorsk
  - The Federal State Budgetary Healthcare Institution The Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - Federal State Institution "Polyclinic No. 5" of the Administrative Department of the President of the Russian Federation, Moscow
  - Podolskaya City Clinical Hospital No. 3, Podolsk
  - Central City Clinical Hospital of Reutov, Reutov
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 25", Saint Petersburg
  - St. Petersburg State Health Care Institution "City Polyclinic №117", Saint Petersburg
  - Road Clinical Hospital JSC Russian Railways, Saint Petersburg
  - LLC "Research Center Eco-Security", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 51", Saint Petersburg
  - St. Petersburg City State Hospital "City Hospital No. 26", Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health "City Polyclinic №34", Saint Petersburg
  - Saratov City Clinical Hospital № 2 named after VI Razumovsky, Saratov
  - Regional State Budgetary Healthcare Institution "Clinical Hospital No.1", Smolensk
  - Yaroslavl State Medical University, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Anaferon: 1 tablet per administration. Day 1: 1 tablet every 30 minutes for the first 2 hours, followed by 3 more tablets taken at regular intervals through the rest of the day.
  Days 2-5: 1 tablet 3 times a day. The drug is taken out of the meal (in the interval between meals or 15-30 minutes before eating), keep the tablet in the mouth, without swallowing, until completely dissolved.
  Anaferon: Oral administration.
Period: Overall Study
Arm/Group | Anaferon | Placebo
Started | 104 | 100
Completed | 103 | 100
Not Completed | 1 | 0
Not completed — Violation of inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaferon | Placebo | Total
Number analyzed (Participants) | 103 | 100 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 100 | 203
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.4) | 37.8 (11.9) | 38.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 139
  Male | 37 | 27 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 103 | 100 | 203

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Acute Respiratory Viral Infection (ARVI) Symptoms.
Description: Based on a patient diary. ARVI is clinically diagnosed and/or Real-time reverse transcription polymerase chain reaction (PCR) confirmed. Criteria of resolution of ARVI symptoms: body/axillary temperature ≤37.30С for 24 hours (without subsequent increase within the observation period) + absence/presence of general ARVI symptoms with ≤2 points of Total Severity (TS) score according to the 4-point scale for each of 14 ARVI symptoms (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). ARVI symptoms are body temperature, 6 nonspecific/flu-like symptoms, and 7 nasal/throat and chest symptoms. Absolute body temperature (in degrees Celsius) is converted to arbitrary units (or scores) using the following scale:
  ≤37.30С=0 points; 37.4-38.00С=1 point; 38.1-39.00С=2 points; ≥39.10С=3 points. TS ranges from 0 to 42 (higher scores mean a worse outcome).
Time Frame: On days 1-7 of the observation period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 103 | 100
days | 4.1 (1.6) | 4.5 (1.5)
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: ARVI Severity.
Description: ARVI severity is assessed using the "Area under the curve" (AUC) for the Total Symptom (TS) score for 6 days of the treatment and observation. TS score is calculated every day according to the 4-point scale for each of 14 ARVI symptoms (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). ARVI symptoms are body temperature, 6 nonspecific/flu-like symptoms, and 7 nasal/throat and chest symptoms. Absolute body temperature (in degrees Celsius) is converted to arbitrary units (or scores) using the following scale: ≤37.30С=0 points; 37.4-38.00С=1 point; 38.1-39.00С=2 points; ≥39.10С=3 points. TS ranges from 0 to 42 (higher scores mean a worse outcome). AUC is calculated between 6 points (by TS for every 6 days of the treatment and observation). AUC is calculated using integration with given limits (TS score). The minimum value for the AUC is "0" and the maximum value is "252" units (day*score). The higher score means a worse outcome (ARVI severity).
Time Frame: On days 1-6 of the observation period.
Measure: Mean (Standard Deviation); unit: day*score
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 103 | 100
day*score | 104.6 (43.5) | 114.3 (45.7)
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Patients With Resolution of ARVI Symptoms (Clinically Diagnosed and/or PCR-confirmed).
Description: Based on patient diary data. Criteria of resolution of ARVI symptoms: body/axillary temperature ≤37.30С for 24 hours (without subsequent increase within the observation period) + absence/presence of general ARVI symptoms with ≤2 points of Total Severity (TS) score according to the 4-point scale for each of 14 ARVI symptoms (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). ARVI symptoms are body temperature, 6 nonspecific/flu-like symptoms, and 7 nasal/throat and chest symptoms. Absolute body temperature (in degrees Celsius) is converted to arbitrary units (or scores) using the following scale: ≤37.30С=0 points; 37.4-38.00С=1 point; 38.1-39.00С=2 points; ≥39.10С=3 points. TS ranges from 0 to 30 (higher scores mean a worse outcome).
Time Frame: On day 2, 3, 4, 5, and 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 103 | 100
Participants
  Day 2 | 0 | 0
  Day 3 | 11 | 6
  Day 4 | 39 | 25
  Day 5 | 57 | 43
  Day 6 | 76 | 64
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Anaferon vs Placebo; Test type: Other — Test for assessing the homogeneity of the odds ratio in several 2 × 2 contingency tables; p = 0.98, Breslow-Day test

4. Secondary Outcome: Time to Resolution of ARVI (PCR-confirmed) Symptoms.
Description: Based on patient diary data. Criteria of resolution of ARVI symptoms: body/axillary temperature ≤37.30С for 24 hours (without subsequent increase within the observation period) + absence/presence of general ARVI symptoms with ≤2 points of Total Severity (TS) score according to the 4-point scale for each of 14 ARVI symptoms (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). ARVI symptoms are body temperature, 6 nonspecific/flu-like symptoms, and 7 nasal/throat and chest symptoms. Absolute body temperature (in degrees Celsius) is converted to arbitrary units (or scores) using the following scale: ≤37.30С=0 points; 37.4-38.00С=1 point; 38.1-39.00С=2 points; ≥39.10С=3 points. TS ranges from 0 to 42 (higher scores mean a worse outcome).
Time Frame: On days 2-6 of the observation period.
Population: From all patients with ARVI only 79 have ARVI (PCR-confirmed), including 41 patient in Anaferon group and 38 patient in Placebo groupe.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 41 | 38
days | 3.6 (1.5) | 4.6 (1.5)
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Patients With Resolution of ARVI Symptoms (PCR-confirmed).
Description: Based on patient diary data. ARVI is PCR confirmed. Criteria of resolution of ARVI symptoms: body/axillary temperature ≤37.30С for 24 hours (without subsequent increase within the observation period) + absence/presence of general ARVI symptoms with ≤2 points of Total Severity (TS) score according to the 4-point scale for each of 14 ARVI symptoms (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). ARVI symptoms are body temperature, 6 nonspecific/flu-like symptoms, and 7 nasal/throat and chest symptoms. Absolute body temperature (in degrees Celsius) is converted to arbitrary units (or scores) using the following scale: ≤37.30С=0 points; 37.4-38.00С=1 point; 38.1-39.00С=2 points; ≥39.10С=3 points. TS ranges from 0 to 30 (higher scores mean a worse outcome).
Time Frame: On day 2, 3, 4, 5, and 6.
Population: From all patients with ARVI only 79 have ARVI (PCR-confirmed), including 41 patient in Anaferon group and 38 patient in Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 41 | 38
Participants
  Day 2 | 0 | 0
  Day 3 | 7 | 4
  Day 4 | 22 | 10
  Day 5 | 29 | 14
  Day 6 | 35 | 23
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Anaferon vs Placebo; Test type: Other — Test for assessing the homogeneity of the odds ratio in several 2 × 2 contingency tables; p = 0.75, Breslow-Day test

6. Secondary Outcome: Dosing Frequency of Antipyretics if Indicated.
Description: Based on patient diary data. Dosing frequency is calculated as the number of antipyretic doses per 1 patient in a day.
Time Frame: On day 1, 2, and 3.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 103 | 100
doses
  Day 1 | 0.4 (0.6) | 0.4 (0.6)
  Day 2 | 0.2 (0.4) | 0.2 (0.4)
  Day 3 | 0.1 (0.3) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Day 1 comparison; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Anaferon vs Placebo; Day 2 comparison; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Anaferon vs Placebo; Day 3 comparison; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: The Percentage of Patients Requiring Administration of Antibiotics.
Description: Based on medical records. This Outcome Measure is calculated as the number of patients who were administered antibiotics for the treatment of secondary bacterial complications.
Time Frame: On days 4-7 of the observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon | Placebo
Number analyzed (Participants) | 103 | 100
Participants | 4 | 5
Statistical Analysis 1: Comparison: Anaferon vs Placebo; Test type: Superiority; p = 0.75, Fisher Exact

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Anaferon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/100
Other Adverse Events (participants affected / at risk) | 5/104 | 5/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon (N=104) | Placebo (N=100)
Intoxication Syndrome Intensification (General disorders) | 0 (0) | 1 (1)
Community-acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acute tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Community-acquired bacterial infection with bacterial bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Community-acquired bacterial infection with purulent rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Acute tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03707912/Prot_SAP_000.pdf